CLINICAL TRIAL: NCT04868968
Title: An Open-label, Single Arm Phase II Study of DFV890 to Assess the Safety, Tolerability and Efficacy in Participants With Familial Cold Auto-inflammatory Syndrome (FCAS)
Brief Title: Study of Safety, Tolerability and Efficacy of DFV890 in Participants With Familial Cold Auto-inflammatory Syndrome (FCAS)
Acronym: DFV890-FCAS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDFV890A12201; 2020-005948-33 (EudraCT Number)
Record Dates: First submitted 2021-04-22; First posted 2021-05-03 (Actual); Results first posted 2024-05-03 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Familial Cold Autoinflammatory Syndrome
Keywords: Familial Cold Auto-inflammatory Syndrome; FCAS; DFV890; NLRP3 inhibitor, inflammasome inhibition; Cryopyrin-associated periodic syndromes; CAPS
MeSH Terms: conditions — Cryopyrin-Associated Periodic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- DFV890 (Experimental): DFV890
  Interventions: Drug: DFV890

INTERVENTIONS:
Drug: DFV890 — 100 mg of DFV890 film coated tablets twice daily (b.i.d.). for 3 days starting in the morning of Day 1 and 100 mg of DFV890 in the morning on the fourth day.

SUMMARY:
The purpose of this phase II study was to assess the safety, tolerability and efficacy of DFV890 in participants with FCAS.

DETAILED DESCRIPTION:
This was an open-label, single-arm, multiple dose, phase II study to assess safety, tolerability and clinical efficacy of DFV890 in participants with FCAS who showed evidence of inflammatory activity after the cold challenge performed during screening.

The study included a screening period, a treatment period and a follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained before any study-specific assessment is performed
* Body mass index within the range of 18-35 kg/m2
* Patients with a genetic diagnosis of FCAS
* Patients with a clinical history and investigations consistent with FCAS

Exclusion Criteria:

* Anti-rejection and/or immunomodulatory drugs must be discontinued (please, see protocol for further details)
* Clinically significant, suspected active or chronic bacterial (including Mycobacterium tuberculosis), viral or fungal infection within 30 days prior to Day 1.
* Patients with innate (e.g. TLR immunodeficiencies, defects in IFN-γ signaling) or acquired immune deficiencies (e.g. AIDS).
* Presence of human immunodeficiency virus (HIV) infection, hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (anti-HBc), or hepatitis C antibodies at screening.
* Live vaccines within 4 weeks of Day 1
* Pregnant or nursing (lactating) women.
* Women of child-bearing potential unless they are using highly effective methods of contraception.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2022-12-13 (Actual); Study Completion 2023-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (3):
- Novartis Investigative Site, La Jolla, California, United States
- Novartis Investigative Site, Paris, France
- Novartis Investigative Site, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1980

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in 3 investigative sites in 3 countries.
Pre-assignment Details: During the screening period the participant's eligibility was assessed at a screening visit and a screening cold challenge was performed.
Groups:
- DFV890 100mg - Treatment: DFV890 100mg oral dose, twice daily for 3 days and one last dose in the morning of Day 4 of the treatment period
Period: Overall Study
Arm/Group | DFV890 100mg - Treatment
Started (All participants enrolled in the trial) | 4
Completed | 3
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | DFV890 100mg - Treatment
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.3 (15.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  other | 1
  white | 3

OUTCOME MEASURES:

1. Primary Outcome: Ratio of Fold Change From Pre-challenge to the Highest Post-challenge Value of White Cell Count (WCC) Between Treatment and Screening Period
Description: A cold challenge was performed during the screening period and on Day 4 of the treatment period. Fold change from pre-challenge to highest post-challenge value of WCC was defined as the ratio of the highest post-challenge WCC value to the pre-challenge WCC value. The ratio of fold change was defined as treatment fold change divided by the screen fold change. A value of less than 1 for the ratio of fold change indicates a lower relative increase of WCC in the treatment than in the screening period, which is a favorable outcome. The log-transformed fold change from pre-challenge to the highest post challenge WCC was analyzed using a log-linear mixed effect model. The analysis was carried out considering the data from -2 to 8 hrs post challenge. The unforeseen screen failure rate and recruitment challenges resulted in early closure of the study. Only 4 out of planned 6 participants were enrolled in the study; thus, the results should be interpreted cautiously.
Time Frame: Screening period and treatment period (Day 4): pre cold challenge and up to 8 hours post cold challenge. The duration of the cold challenge was 45 minutes.
Population: The Pharmacodynamic (PD) analysis set included all participants with no protocol deviations with relevant impact on PD data.
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: ratio of fold change
Groups:
- DFV890 100mg: DFV890 100mg oral dose, twice daily for 3 days and one last dose in the morning of Day 4 of the treatment period
Arm/Group | DFV890 100mg
Number analyzed (Participants) | 4
ratio of fold change | 0.82 [0.56 to 1.21]

2. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Number of participants with treatment emergent AEs (any AE regardless of seriousness), AEs led to study treatment discontinuation, SAEs and SAEs led to study treatment discontinuation.
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment plus 30 days post treatment, up to a maximum duration of approximately 34 days
Population: The safety analysis set included all participants that received any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | DFV890 100mg - Treatment
Number analyzed (Participants) | 4
Participants
  At least one AE | 4
  At least one SAE | 0
  AE leading to discontinuation | 0
  SAE leading to discontinuation | 0

3. Secondary Outcome: Physician Global Assessment of Autoinflammatory Disease Activity
Description: The Physician global assessment of autoinflammatory disease activity is a questionnaire completed by the Investigator. It uses a 5-point scale. Lower scores represent better outcomes.
  0 = Absent
  1. = Minimal
  2. = Mild
  3. = Moderate
  4. = Severe
Time Frame: Screening and Treatment (Day 4): 1 hour pre and 2, 3, 5, 9 and 24 hours post. Scheduled time refers to the time post-meal (screening) and to the time post-dose (treatment). The start of the cold challenge is at 1 hour post and the duration is 45 minutes.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Screening: Screening period
Arm/Group | Screening | DFV890 100mg - Treatment
Number analyzed (Participants) | 4 | 4
Participants
  1 hour pre: Absent | 0 | 2
  1 hour pre: Minimal | 3 | 2
  1 hour pre: Mild | 1 | 0
  1 hour pre: Moderate | 0 | 0
  1 hour pre: Severe | 0 | 0
  2 hours post: Absent | 0 | 2
  2 hours post: Minimal | 2 | 1
  2 hours post: Mild | 2 | 1
  2 hours post: Moderate | 0 | 0
  2 hours post: Severe | 0 | 0
  3 hours post: Absent | 0 | 2
  3 hours post: Minimal | 1 | 1
  3 hours post: Mild | 3 | 1
  3 hours post: Moderate | 0 | 0
  3 hours post: Severe | 0 | 0
  5 hours post: Absent | 0 | 2
  5 hours post: Minimal | 1 | 1
  5 hours post: Mild | 3 | 1
  5 hours post: Moderate | 0 | 0
  5 hours post: Severe | 0 | 0
  9 hours post: Absent | 0 | 1
  9 hours post: Minimal | 1 | 2
  9 hours post: Mild | 0 | 1
  9 hours post: Moderate | 3 | 0
  9 hours post: Severe | 0 | 0
  24 hours post: Absent | 0 | 2
  24 hours post: Minimal | 3 | 2
  24 hours post: Mild | 1 | 0
  24 hours post: Moderate | 0 | 0
  24 hours post: Severe | 0 | 0

4. Secondary Outcome: Physician's Severity Assessment of Autoinflammatory Disease Signs and Symptoms
Description: The Physician's severity assessment of autoinflammatory disease signs and symptoms is a questionnaire completed by the Investigator. It uses a 5-point scale. Lower scores represent better outcomes.
  0 = Absent
  1. = Minimal
  2. = Mild
  3. = Moderate
  4. = Severe
  The following items were assessed:
  * Assessment of skin disease (urticarial skin rash)
  * Assessment of arthralgia
  * Assessment of myalgia
  * Assessment of headache/migraine
  * Assessment of conjunctivitis
  * Assessment of fatigue/malaise
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Screening | DFV890 100mg - Treatment
Number analyzed (Participants) | 4 | 4
Participants
  Arthralgia 1 hour pre: Absent | 3 | 3
  Arthralgia 1 hour pre: Minimal | 1 | 1
  Arthralgia 1 hour pre: Mild | 0 | 0
  Arthralgia 1 hour pre: Moderate | 0 | 0
  Arthralgia 1 hour pre: Severe | 0 | 0
  Arthralgia 2 hours post: Absent | 4 | 4
  Arthralgia 2 hours post: Minimal | 0 | 0
  Arthralgia 2 hours post: Mild | 0 | 0
  Arthralgia 2 hours post: Moderate | 0 | 0
  Arthralgia 2 hours post: Severe | 0 | 0
  Arthralgia 3 hours post: Absent | 4 | 4
  Arthralgia 3 hours post: Minimal | 0 | 0
  Arthralgia 3 hours post: Mild | 0 | 0
  Arthralgia 3 hours post: Moderate | 0 | 0
  Arthralgia 3 hours post: Severe | 0 | 0
  Arthralgia 5 hours post: Absent | 3 | 4
  Arthralgia 5 hours post: Minimal | 0 | 0
  Arthralgia 5 hours post: Mild | 1 | 0
  Arthralgia 5 hours post: Moderate | 0 | 0
  Arthralgia 5 hours post: Severe | 0 | 0
  Arthralgia 9 hours post: Absent | 1 | 3
  Arthralgia 9 hours post: Minimal | 3 | 1
  Arthralgia 9 hours post: Mild | 0 | 0
  Arthralgia 9 hours post: Moderate | 0 | 0
  Arthralgia 9 hours post: Severe | 0 | 0
  Arthralgia 24 hours post: Absent | 4 | 3
  Arthralgia 24 hours post: Minimal | 0 | 1
  Arthralgia 24 hours post: Mild | 0 | 0
  Arthralgia 24 hours post: Moderate | 0 | 0
  Arthralgia 24 hours post: Severe | 0 | 0
  Conjunctivitis 1 hour pre: Absent | 3 | 3
  Conjunctivitis 1 hour pre: Minimal | 0 | 1
  Conjunctivitis 1 hour pre: Mild | 1 | 0
  Conjunctivitis 1 hour pre: Moderate | 0 | 0
  Conjunctivitis 1 hour pre: Severe | 0 | 0
  Conjunctivitis 2 hours post: Absent | 3 | 4
  Conjunctivitis 2 hours post: Minimal | 0 | 0
  Conjunctivitis 2 hours post: Mild | 1 | 0
  Conjunctivitis 2 hours post: Moderate | 0 | 0
  Conjunctivitis 2 hours post: Severe | 0 | 0
  Conjunctivitis 3 hours post: Absent | 3 | 4
  Conjunctivitis 3 hours post: Minimal | 0 | 0
  Conjunctivitis 3 hours post: Mild | 1 | 0
  Conjunctivitis 3 hours post: Moderate | 0 | 0
  Conjunctivitis 3 hours post: Severe | 0 | 0
  Conjunctivitis 5 hours post: Absent | 3 | 4
  Conjunctivitis 5 hours post: Minimal | 0 | 0
  Conjunctivitis 5 hours post: Mild | 1 | 0
  Conjunctivitis 5 hours post: Moderate | 0 | 0
  Conjunctivitis 5 hours post: Severe | 0 | 0
  Conjunctivitis 9 hours post: Absent | 2 | 4
  Conjunctivitis 9 hours post: Minimal | 0 | 0
  Conjunctivitis 9 hours post: Mild | 1 | 0
  Conjunctivitis 9 hours post: Moderate | 1 | 0
  Conjunctivitis 9 hours post: Severe | 0 | 0
  Conjunctivitis 24 hours post: Absent | 3 | 2
  Conjunctivitis 24 hours post: Minimal | 0 | 2
  Conjunctivitis 24 hours post: Mild | 1 | 0
  Conjunctivitis 24 hours post: Moderate | 0 | 0
  Conjunctivitis 24 hours post: Severe | 0 | 0
  Fatigue/Malaise 1 hour pre: Absent | 3 | 3
  Fatigue/Malaise 1 hour pre: Minimal | 0 | 0
  Fatigue/Malaise 1 hour pre: Mild | 1 | 1
  Fatigue/Malaise 1 hour pre: Moderate | 0 | 0
  Fatigue/Malaise 1 hour pre: Severe | 0 | 0
  Fatigue/Malaise 2 hours post: Absent | 3 | 3
  Fatigue/Malaise 2 hours post: Minimal | 0 | 0
  Fatigue/Malaise 2 hours post: Mild | 1 | 0
  Fatigue/Malaise 2 hours post: Moderate | 0 | 1
  Fatigue/Malaise 2 hours post: Severe | 0 | 0
  Fatigue/Malaise 3 hours post: Absent | 2 | 3
  Fatigue/Malaise 3 hours post: Minimal | 1 | 0
  Fatigue/Malaise 3 hours post: Mild | 0 | 0
  Fatigue/Malaise 3 hours post: Moderate | 1 | 1
  Fatigue/Malaise 3 hours post: Severe | 0 | 0
  Fatigue/Malaise 5 hours post: Absent | 2 | 3
  Fatigue/Malaise 5 hours post: Minimal | 0 | 0
  Fatigue/Malaise 5 hours post: Mild | 2 | 0
  Fatigue/Malaise 5 hours post: Moderate | 0 | 1
  Fatigue/Malaise 5 hours post: Severe | 0 | 0
  Fatigue/Malaise 9 hours post: Absent | 2 | 3
  Fatigue/Malaise 9 hours post: Minimal | 0 | 0
  Fatigue/Malaise 9 hours post: Mild | 1 | 0
  Fatigue/Malaise 9 hours post: Moderate | 1 | 1
  Fatigue/Malaise 9 hours post: Severe | 0 | 0
  Fatigue/Malaise 24 hours post: Absent | 3 | 3
  Fatigue/Malaise 24 hours post: Minimal | 1 | 1
  Fatigue/Malaise 24 hours post: Mild | 0 | 0
  Fatigue/Malaise 24 hours post: Moderate | 0 | 0
  Fatigue/Malaise 24 hours post: Severe | 0 | 0
  Headache/Migraine 1 hour pre: Absent | 4 | 4
  Headache/Migraine 1 hour pre: Minimal | 0 | 0
  Headache/Migraine 1 hour pre: Mild | 0 | 0
  Headache/Migraine 1 hour pre: Moderate | 0 | 0
  Headache/Migraine 1 hour pre: Severe | 0 | 0
  Headache/Migraine 2 hours post: Absent | 4 | 4
  Headache/Migraine 2 hours post: Minimal | 0 | 0
  Headache/Migraine 2 hours post: Mild | 0 | 0
  Headache/Migraine 2 hours post: Moderate | 0 | 0
  Headache/Migraine 2 hours post: Severe | 0 | 0
  Headache/Migraine 3 hours post: Absent | 4 | 4
  Headache/Migraine 3 hours post: Minimal | 0 | 0
  Headache/Migraine 3 hours post: Mild | 0 | 0
  Headache/Migraine 3 hours post: Moderate | 0 | 0
  Headache/Migraine 3 hours post: Severe | 0 | 0
  Headache/Migraine 5 hours post: Absent | 4 | 4
  Headache/Migraine 5 hours post: Minimal | 0 | 0
  Headache/Migraine 5 hours post: Mild | 0 | 0
  Headache/Migraine 5 hours post: Moderate | 0 | 0
  Headache/Migraine 5 hours post: Severe | 0 | 0
  Headache/Migraine 9 hours post: Absent | 3 | 4
  Headache/Migraine 9 hours post: Minimal | 0 | 0
  Headache/Migraine 9 hours post: Mild | 1 | 0
  Headache/Migraine 9 hours post: Moderate | 0 | 0
  Headache/Migraine 9 hours post: Severe | 0 | 0
  Headache/Migraine 24 hours post: Absent | 4 | 4
  Headache/Migraine 24 hours post: Minimal | 0 | 0
  Headache/Migraine 24 hours post: Mild | 0 | 0
  Headache/Migraine 24 hours post: Moderate | 0 | 0
  Headache/Migraine 24 hours post: Severe | 0 | 0
  Myalgia 1 hour pre: Absent | 3 | 4
  Myalgia 1 hour pre: Minimal | 1 | 0
  Myalgia 1 hour pre: Mild | 0 | 0
  Myalgia 1 hour pre: Moderate | 0 | 0
  Myalgia 1 hour pre: Severe | 0 | 0
  Myalgia 2 hours post: Absent | 4 | 3
  Myalgia 2 hours post: Minimal | 0 | 1
  Myalgia 2 hours post: Mild | 0 | 0
  Myalgia 2 hours post: Moderate | 0 | 0
  Myalgia 2 hours post: Severe | 0 | 0
  Myalgia 3 hours post: Absent | 3 | 4
  Myalgia 3 hours post: Minimal | 0 | 0
  Myalgia 3 hours post: Mild | 1 | 0
  Myalgia 3 hours post: Moderate | 0 | 0
  Myalgia 3 hours post: Severe | 0 | 0
  Myalgia 5 hours post: Absent | 3 | 4
  Myalgia 5 hours post: Minimal | 0 | 0
  Myalgia 5 hours post: Mild | 1 | 0
  Myalgia 5 hours post: Moderate | 0 | 0
  Myalgia 5 hours post: Severe | 0 | 0
  Myalgia 9 hours post: Absent | 3 | 4
  Myalgia 9 hours post: Minimal | 1 | 0
  Myalgia 9 hours post: Mild | 0 | 0
  Myalgia 9 hours post: Moderate | 0 | 0
  Myalgia 9 hours post: Severe | 0 | 0
  Myalgia 24 hours post: Absent | 4 | 4
  Myalgia 24 hours post: Minimal | 0 | 0
  Myalgia 24 hours post: Mild | 0 | 0
  Myalgia 24 hours post: Moderate | 0 | 0
  Myalgia 24 hours post: Severe | 0 | 0
  Skin disease 1 hour pre: Absent | 0 | 1
  Skin disease 1 hour pre: Minimal | 3 | 3
  Skin disease 1 hour pre: Mild | 1 | 0
  Skin disease 1 hour pre: Moderate | 0 | 0
  Skin disease 1 hour pre: Severe | 0 | 0
  Skin disease 2 hours post: Absent | 0 | 1
  Skin disease 2 hours post: Minimal | 2 | 3
  Skin disease 2 hours post: Mild | 2 | 0
  Skin disease 2 hours post: Moderate | 0 | 0
  Skin disease 2 hours post: Severe | 0 | 0
  Skin disease 3 hours post: Absent | 0 | 2
  Skin disease 3 hours post: Minimal | 1 | 2
  Skin disease 3 hours post: Mild | 3 | 0
  Skin disease 3 hours post: Moderate | 0 | 0
  Skin disease 3 hours post: Severe | 0 | 0
  Skin disease 5 hours post: Absent | 0 | 2
  Skin disease 5 hours post: Minimal | 1 | 2
  Skin disease 5 hours post: Mild | 3 | 0
  Skin disease 5 hours post: Moderate | 0 | 0
  Skin disease 5 hours post: Severe | 0 | 0
  Skin disease 9 hours post: Absent | 0 | 1
  Skin disease 9 hours post: Minimal | 1 | 3
  Skin disease 9 hours post: Mild | 0 | 0
  Skin disease 9 hours post: Moderate | 3 | 0
  Skin disease 9 hours post: Severe | 0 | 0
  Skin disease 24 hours post: Absent | 0 | 2
  Skin disease 24 hours post: Minimal | 3 | 2
  Skin disease 24 hours post: Mild | 1 | 0
  Skin disease 24 hours post: Moderate | 0 | 0
  Skin disease 24 hours post: Severe | 0 | 0

5. Secondary Outcome: Patient's Global Assessment of Disease Activity
Description: Patient's global assessment of disease activity is a questionnaire completed by the patient. It uses a 5-point scale. The patient selected a rating based on the patient's current disease activity at the time of the assessment. Lower scores represent better outcomes.
  0 = Absent
  1. = Minimal
  2. = Mild
  3. = Moderate
  4. = Severe
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Screening | DFV890 100mg - Treatment
Number analyzed (Participants) | 4 | 4
Participants
  1 hour pre: Absent | 2 | 3
  1 hour pre: Minimal | 2 | 1
  1 hour pre: Mild | 0 | 0
  1 hour pre: Moderate | 0 | 0
  1 hour pre: Severe | 0 | 0
  2 hours post: Absent | 0 | 3
  2 hours post: Minimal | 4 | 0
  2 hours post: Mild | 0 | 1
  2 hours post: Moderate | 0 | 0
  2 hours post: Severe | 0 | 0
  3 hours post: Absent | 0 | 3
  3 hours post: Minimal | 2 | 0
  3 hours post: Mild | 2 | 1
  3 hours post: Moderate | 0 | 0
  3 hours post: Severe | 0 | 0
  5 hours post: Absent | 0 | 2
  5 hours post: Minimal | 2 | 2
  5 hours post: Mild | 2 | 0
  5 hours post: Moderate | 0 | 0
  5 hours post: Severe | 0 | 0
  9 hours post: Absent | 0 | 2
  9 hours post: Minimal | 1 | 2
  9 hours post: Mild | 2 | 0
  9 hours post: Moderate | 1 | 0
  9 hours post: Severe | 0 | 0
  24 hours post: Absent | 1 | 2
  24 hours post: Minimal | 3 | 2
  24 hours post: Mild | 0 | 0
  24 hours post: Moderate | 0 | 0
  24 hours post: Severe | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment plus 30 days post treatment, up to a maximum duration of approximately 34 days
Groups:
- DFV890 100 mg - Treatment: DFV890 100mg oral dose, twice daily for 3 days and one last dose in the morning of Day 4 of the treatment period
Arm/Group | DFV890 100 mg - Treatment
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 4/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DFV890 100 mg - Treatment (N=4)
Asthenia (General disorders) | 1
Chills (General disorders) | 1
Fatigue (General disorders) | 2
Conjunctivitis (Infections and infestations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Cold urticaria (Skin and subcutaneous tissue disorders) | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-05-19): https://cdn.clinicaltrials.gov/large-docs/68/NCT04868968/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-17): https://cdn.clinicaltrials.gov/large-docs/68/NCT04868968/SAP_001.pdf